CLINICAL TRIAL: NCT00837681
Title: Pulmonary Complications of Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Karen Wood (Other)
Responsible Party: Sponsor-Investigator, Karen Wood, Karen Wood M.D., Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2005C0058
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2016-07

CONDITIONS: Lung Disease
Keywords: Bone Marrow Transplant; hematopoietic stem cell transplantation
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw will be 10cc of blood, analysis includes % of CD8+CD57+ and CD8+CD28-. On one occasion, after the 6 mo. post transplant timepoint the subject will be asked to donate a larger amount of blood (50cc) if they are not anemic.
  ***Respiratory Specimens of extra BAL or biopsy specimens will be collected at any point a study patient undergoes a clinically warranted bronchoscopy or lung biopsy procedure and the diagnostic physician feels there is adequate specimen to use extra sample for research purposes.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lung disease: hematopoietic stem cell transplantation (HSCT)

SUMMARY:
The purpose of this study is to determine risk factors associated with the development of lung disease after hematopoietic stem cell transplantation. Depending on the results and findings of this study, it may be possible to predict who is at higher risk of serious complications and ultimately develop therapies to prevent or treat this lung disease.

DETAILED DESCRIPTION:
The development of pulmonary complications after hematopoietic stem cell transplantation is responsible for significant morbidity and mortality. The incidence of pulmonary disease has been reported to be as high as 50% of all patients that undergo transplant. The most common manifestation of early onset lung disease is idiopathic pneumonia syndrome. This can occur in autologous and allogeneic transplants, with an incidence between 5% and 10% and a mortality rate as high as 74%(1). Late onset pulmonary disease may be even more frequent and has been reported between 10-24% in recipients of allogeneic HSCT(2-4). Additionally, a recent study demonstrated 26% of patients develop airflow obstruction after transplant and this was correlated with mortality(5). One quite useful classification system divides late onset pulmonary disease into bronchiolitis obliterans and interstitial pneumonia(4). Interstitial pneumonia is a condition characterized by diffuse infiltrates, often with lymphocyte predominance, and associated with restrictive defects on pulmonary function testing. Bronchiolitis obliterans is characterized by progressive airflow obstruction and a normal radiograph (except possibly associated air trapping). The incidence of bronchiolitis obliterans after HSCT varies widely, but is usually reported to be between 1% and 11%(6-8), although the presence of post HSCT obstructive airway disease was reported at 26% in a recent large study(5). Late onset pulmonary diseases are often treated with increased immunosuppression, but the prognosis is poor with limited response to therapy(9; 4).

ELIGIBILITY:
Inclusion Criteria:

1. All patients scheduled to undergo hematopoietic stem cell transplantation (HSCT)

Exclusion Criteria:

1. Patients whose ability to give informed consent is in question.
2. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled to undergo hematopoietic stem cell transplantation (HSCT)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2005-10; Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

PRIMARY OUTCOMES:
To determine factors contributing to the development of lung disease after hematopoietic stem cell transplantation (HSCT | end of study

SECONDARY OUTCOMES:
1b) To identify the mechanisms by which CD8+ regulatory cells suppress the alloimmune response. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wood, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States